CLINICAL TRIAL: NCT00984542
Title: Phase II Study of Second-Line Bendamustine in Relapsed or Refractory Small Cell Lung Cancer (SCLC).
Brief Title: Bendamustine as Second-Line Therapy in Treating Patients With Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Leora Horn, MD, Assistant Professor of Medicine; Assistant Director, Educator Development Program; Clinical Director, Thoracic Oncology Program; Medical Oncologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC THO 0920; P30CA068485 (NIH); VU-VICC-THO-0920
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2014-03-12 (Estimated); Last update posted 2014-03-12 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer
Keywords: recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bendamustine (Experimental)
  Interventions: Drug: bendamustine hydrochloride

INTERVENTIONS:
Drug: bendamustine hydrochloride — Bendamustine 120 mg/m2 IV on days 1 and 2 of a 21-day treatment cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as bendamustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well bendamustine works as second- or third-line therapy in treating patients with relapsed or refractory small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the time to progression in patients with relapsed or refractory small cell lung cancer treated with second- or third-line bendamustine.

Secondary

* To determine the toxicity of this drug in these patients.
* To determine the response rate, progression-free survival, and overall survival of patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive bendamustine IV over 1 hour on days 1 and 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6-8 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed small cell lung cancer
* Relapsed or refractory disease after 1-2 prior chemotherapy regimens
* Measurable disease
* ECOG - Eastern Cooperative Oncology Group performance status 0-2
* ANC ≥ 1,500/mm³: ANC = Absolute neutrophil count
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 9 g/dL
* Bilirubin normal
* AST/ALT ≤ 2 times upper limit of normal (ULN) (≤ 5 times ULN in patients with hepatic metastases; AST/ALT = alanine transaminase (ALT) and aspartate aminotransferase (AST)
* Creatinine clearance > 40 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception before, during, and for ≥ 3 months after completion of study therapy
* No known hypersensitivity to bendamustine
* No other malignancy for which the patient has been treated within the past year except for nonmelanoma skin cancer or carcinoma in situ of the cervix
* No cardiac disease, including any of the following:

  * Unstable angina pectoris
  * Life-threatening cardiac arrhythmia
  * Symptomatic congestive heart failure
* No uncontrolled infection
* No other concurrent chemotherapy, immunotherapy, or anti-tumor hormonal therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leora Horn, M.D., Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (6):
- United States (6):
  - Hardin Memorial Hosptial, Elizabethtown, Kentucky
  - The Jones Clinic - Germantown, Germantown, Tennessee
  - Jackson-Madison County Hospital, Jackson, Tennessee
  - Baptist Regional Cancer Center at Baptist Riverside, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study opened to accrual in September 2009 and closed to accrual in February 2012
Pre-assignment Details: 59 patients consented, 9 were determined to be ineligible to participate
Groups:
- Bendamustine: Bendamustine 120 mg/m2 of body surface area intravenously on days 1 and 2 of a 21-day treatment cycle for a maximum of six cycles
Period: Overall Study
Arm/Group | Bendamustine
Started | 50
Completed | 9
Not Completed | 41
Not completed — disease progression | 19
Not completed — toxicity | 7
Not completed — Death | 7
Not completed — complicating disease | 3
Not completed — Withdrawal by Subject | 3
Not completed — clinical deterioration | 2

BASELINE CHARACTERISTICS:
Population: Patients with Relapsed or Refractory Small Cell Lung Cancer (SCLC)who received study drug
Arm/Group | Bendamustine
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Time to Progression
Description: Estimated probable duration from on-study date to date of disease progression, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: On-study to date of progression, measured following cycle 2, 4, and 6 of a 21-day cycle for 6 cycles, (during 126 days)
Population: All patients are included in the analysis on intention-to treat basis. Analysis is by Kaplan-Meier method, where progression is an event, with censoring for non-progressed patients at greater of off-study date, last known alive date, or date of death not attributable to disease progression.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bendamustine
Number analyzed (Participants) | 50
days | 123 [98 to 138]

2. Secondary Outcome: Number of Patients With Each Worst-grade Toxicity
Description: Number of patients with worst-grade toxicity at each of five grades following NCI Common Toxicity Criteria with grade 1 = mild, grade 2 = moderate, grade 3 = severe, grade 4 = life-threatening/disabling, 5 = death.
Time Frame: Day 1 of each 21-day cycle for 6 cycles and at 30 days after end of treatment, at 156 days
Population: Total number of patients reported with any toxicity
Measure: Number; unit: participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 50
participants
  Number of patients with worst-grade toxicity of 1 | 1
  Number of patients with worst-grade toxicity of 2 | 14
  Number of patients with worst-grade toxicity of 3 | 21
  Number of patients with worst-grade toxicity of 4 | 5
  Number of patients with worst-grade toxicity of 5 | 9

3. Secondary Outcome: Best Response
Description: Number of patients in each response category, per RECIST v1.1, summarized as follows for target lesion criteria (see RECIST v1.1 for additional details):
  complete response (CR),disappearance of target lesions; partial response (PR), >=30% decrease in sum of longest diameter of target lesions; progressive disease (PD), >=20% increase in sum of LD of target lesions or appearance of new lesions; stable disease (SD), insufficient change in target lesions or new lesions to qualify as either PD or SD. Patients are categorized according to the best response achieved prior to occurrence of progressive disease, where best response hierarchy is CR>PR>SD>PD.
Time Frame: On-treatment date to date of disease progression, following cycle 2, 4, and 6 of a 21-day cycle for 6 cycles, (assessed up to 126 days)
Population: All patients with best overall response data; patients are excluded if best overall response data is missing or if the patient is non-evaluable for best overall response. 8 patients were not evaluable.
Measure: Number; unit: participants
Arm/Group | Bendamustine
Number analyzed (Participants) | 42
participants
  Complete Response | 1
  Partial Response | 10
  Progressive Disease | 14
  Stable Disease | 17

4. Secondary Outcome: Progression-free Survival
Description: Estimated probable duration of life without disease progression, from on-study date to earlier of progression date or date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details). Disease progression is defined under RECIST v1.1 as >=20% increase in sum of longest diameters of target lesions, unequivocal progression of non-target lesions, or appearance of new lesions.
Time Frame: On-study date to lesser of date of progression or date of death from any cause ,measured following cycle 2, 4, 6 of a 21-day cycle for 6 cycles, (assessed up to 126 days)
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where either death or progression is an event, with censoring for non-progressed, non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Bendamustine
Number analyzed (Participants) | 50
days | 98 [61 to 114]

5. Secondary Outcome: Overall Survival
Description: Estimated probable duration of life from on-study date to date of death from any cause, using the Kaplan-Meier method with censoring (see analysis population description for additional details)
Time Frame: On study to date of death from any cause or last date known alive, measured every 6-8 weeks from the end of treatment, up to 31 months
Population: All patients are included in the analysis on intention-to-treat basis. Analysis is by Kaplan-Meier method, where death is an event, with censoring for non-expired patients at greater of off-study date or last known alive date.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Bendatmustine: Bendamustine 120 mg/m2 of body surface area intravenously on days 1 and 2 of a 21-day treatment cycle for a maximum of six cycles
Arm/Group | Bendatmustine
Number analyzed (Participants) | 50
days | 144 [110 to 182]

ADVERSE EVENTS:
Arm/Group | Bendamustine
Serious Adverse Events (participants affected / at risk) | 27/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=50)
atrial fibrillation (Cardiac disorders) | 2 (2)
troponin levels postive (Cardiac disorders) | 1 (1)
clot, left upper arm (Vascular disorders) | 1 (1)
chills (General disorders) | 1 (1)
creatine (Investigations) | 1 (1)
death not associated with CTCAE term-NOS (General disorders) | 1 (1)
death not associated with CTCAE term-disease progression (General disorders) | 9 (9)
diarrhea (Gastrointestinal disorders) | 3 (3)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
fatigue (General disorders) | 3 (3)
fever in the absence of neutropenia, where neutropenia is defined as ANC < 1.0 x 10e9/L (General disorders) | 2 (2)
hip fracture (Musculoskeletal and connective tissue disorders) | 3 (3)
glucose, serum-low (Metabolism and nutrition disorders) | 1 (1)
hemoglobin (Blood and lymphatic system disorders) | 3 (3)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
infection-other (Infections and infestations) | 1 (1)
infection-documented with Grade 3 or 4 neutrophils-pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
infection with normal ANC or Grade 1 or 2 neutrophils-bronchus (Respiratory, thoracic and mediastinal disorders) | 1 (1)
infection with normal ANC or Grade 1 or 2 neutrophils-lung (Respiratory, thoracic and mediastinal disorders) | 2 (2)
infection with unknown ANC-lung (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 4 (4)
neutrophils/granulocytes (Blood and lymphatic system disorders) | 2 (2)
pain-abdomen NOS (Gastrointestinal disorders) | 1 (1)
chest pain (Cardiac disorders) | 1 (1)
pain-right hip (Musculoskeletal and connective tissue disorders) | 1 (1)
pain NOS (General disorders) | 1 (1)
pericardial effusion-non-malignant (Cardiac disorders) | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
potassium, serum-low (Metabolism and nutrition disorders) | 1 (1)
acute respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
bilateral basilar pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulomonary emboli-multiple (Respiratory, thoracic and mediastinal disorders) | 1 (1)
right lower lobe lung collapse (Respiratory, thoracic and mediastinal disorders) | 1 (1)
acute renal failure (Renal and urinary disorders) | 1 (1)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
somnolence (Nervous system disorders) | 1 (1)
superior vena cava syndrome (Vascular disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 2 (2)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bendamustine (N=50)
albumin, serum-low (Metabolism and nutrition disorders) | 6 (7)
alkaline phosphatase (Investigations) | 4 (5)
Alanine aminotransferase, serum glutamic pyruvic transaminase (ALT, SGPT) (Investigations) | 4 (5)
anorexia (Metabolism and nutrition disorders) | 16 (20)
aspartate transaminase, serum glutamic oxaloacetic transaminase (AST, SGOT) (Investigations) | 6 (7)
constipation (Gastrointestinal disorders) | 9 (9)
constitutional symptoms-other (General disorders) | 15 (51)
cough (Respiratory, thoracic and mediastinal disorders) | 8 (8)
dermatology/skin-other (Skin and subcutaneous tissue disorders) | 5 (7)
diarrhea (Gastrointestinal disorders) | 9 (13)
dizziness (Nervous system disorders) | 5 (7)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (13)
edema-limb (General disorders) | 4 (4)
fatigue (General disorders) | 25 (39)
calcium, serum-low (Metabolism and nutrition disorders) | 4 (4)
gastrointestinal-other (Gastrointestinal disorders) | 3 (3)
glucose, serum-high (Metabolism and nutrition disorders) | 8 (15)
hemoglobin (Blood and lymphatic system disorders) | 26 (49)
hypotension (Vascular disorders) | 3 (3)
insomnia (Psychiatric disorders) | 5 (5)
leukocytes (Blood and lymphatic system disorders) | 11 (26)
magnesium, serum-low (Metabolism and nutrition disorders) | 5 (8)
metabolic, laboratory-other (Metabolism and nutrition disorders) | 15 (31)
depression (Psychiatric disorders) | 3 (3)
mucositis (functional/symptomatic)-oral cavity (Gastrointestinal disorders) | 3 (3)
nausea (Gastrointestinal disorders) | 21 (24)
neurology-other (Nervous system disorders) | 3 (3)
neuropathy-sensory (Nervous system disorders) | 3 (4)
neutrophils/granulocytes (Blood and lymphatic system disorders) | 6 (9)
pain-abdomen NOS (Gastrointestinal disorders) | 4 (4)
pain-back (Musculoskeletal and connective tissue disorders) | 7 (7)
pain-extremity, limb (Musculoskeletal and connective tissue disorders) | 3 (3)
pain-joint (Musculoskeletal and connective tissue disorders) | 6 (6)
platelets (Blood and lymphatic system disorders) | 17 (31)
potassium, serum-low (Metabolism and nutrition disorders) | 6 (9)
pulmonary/upper respiratory-other (Respiratory, thoracic and mediastinal disorders) | 7 (11)
sodium, serum-low (Investigations) | 9 (14)
vomiting (Gastrointestinal disorders) | 14 (19)
weight loss (Investigations) | 10 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No